CLINICAL TRIAL: NCT06729333
Title: A Multicenter and Prospective Study of Screening Retinopathy of Prematurity in China
Acronym: SChiROP
Status: Not yet recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Peiquan Zhao, Director of the Department of Ophthalmology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-C-2024-205-1
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Premature Birth of Newborn; Retinopathy of Prematurity (ROP); Low Birthweight Infant
Keywords: retinopathy of prematurity; incidence rate; screening
MeSH Terms: conditions — Premature Birth; Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of the study is to explore the current incidence rate of retinopathy of prematurity (ROP) in China and to explore more appropriate screening criteria for ROP.

ELIGIBILITY:
Inclusion Criteria:

From December 2024 to May 2025, preterm infants (gestational age <37 weeks) or low birth weight infants (birth weight <2500 g) who receive their first ROP screening at Xinhua Hospital or partner institutions will be included.

Exclusion Criteria:

1. Death before the first screening;
2. Death or loss to follow-up before complete retinal vascularization;
3. Presence of other diseases causing incomplete retinal vascularization, such as familial exudative vitreoretinopathy, incontinentia pigmenti, or Coats disease;
4. Coexisting conditions affecting the classification or staging of ROP, such as corneal opacity, congenital cataract, persistent fetal vasculature, retinoblastoma, anophthalmia, Terson syndrome, or other ocular infections or diseases;
5. Poor systemic condition preventing fundus examination;
6. History of ocular trauma or surgery (excluding treatments for ROP);
7. Poor-quality fundus images;
8. Other conditions deemed exclusionary by the investigators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-12-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of ROP | 6 months after the first screening
Gestational age at which treatment-requiring ROP develops | 6 months after the first screening
Birthweight at which treatment-requiring ROP develops | 6 months after the first screening

SECONDARY OUTCOMES:
Gestational age of infants developing any ROP lesion | 6 months after the first screening
Birthweight of infants developing any ROP lesion | 6 months after the first screening
Postmenstrual age (PMA) at which ROP lesions occur | 6 months after the first screening
PMA at which treatment-requiring ROP occurs | 6 months after the first screening
Screening and treatment costs | 6 months after the first screening

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China